CLINICAL TRIAL: NCT00896766
Title: Childhood Cancer Therapeutically Applicable Research to Generate Effective Treatments (TARGET) Initiative High-Risk ALL Pilot Project: Application of Array-Based Methods and Gene Re-Sequencing to Identify Candidate Molecular Targets for High-Risk Pediatric Acute Lymphoblastic Leukemia
Brief Title: Laboratory Study of Lymphoblasts in Young Patients With High-Risk Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL06B1; COG-AALL06B1 (Other: Children's Oncology Group); CDR0000496763 (Other: Clinical Trials.gov); NCI-2009-00314 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute lymphoblastic leukemia in remission; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Microarray Analysis; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: loss of heterozygosity analysis
Genetic: microarray analysis
Genetic: polymorphism analysis
Genetic: tumor replication error analysis

SUMMARY:
RATIONALE: Collecting and storing samples of bone marrow and blood from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at lymphoblasts in young patients with high-risk acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify regions of copy number abnormalities (CNA) and uniparental disomy in leukemic lymphoblasts from pediatric patients with high-risk acute lymphoblastic leukemia (ALL) using Affymetrix GeneChip Mapping 500K array sets. (Pilot project)
* Identify regions of CNA and loss-of-heterozygosity using Affymetrix SNP 6.0 microarrays. (Expansion project)
* Define gene expression profiles for leukemic lymphoblasts using Affymetrix U133 Plus 2.0 arrays.
* Assess the global expression of microRNAs in leukemic lymphoblasts using microRNA gene chips.
* Utilize array-generated gene expression data and data for CNAs and uniparental disomy to prioritize candidate genes and genomic regions for resequencing.
* Characterize epigenomic profiles using the HpaII tiny fragment Enrichment by Ligation-mediated PCR (HELP) assay. (Expansion project)
* Discover candidate therapeutic targets for these patients by identifying genes that are consistently mutated in leukemic lymphoblasts using high-throughput focused gene resequencing. (Pilot project)
* Discover candidate therapeutic targets for these patients by next generation sequencing technologies, including whole genome, whole transcriptome, and whole exome. (Expansion project)

OUTLINE: This is a multicenter study.

Banked biological samples (bone marrow and peripheral blood) are analyzed using gene expression profiling, single-nucleotide polymorphism and genotyping assays, DNA copy number and loss of heterozygosity estimates, epigenetic profiling, and gene resequencing.

PROJECTED ACCRUAL: A total of 150 patient samples will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell precursor acute lymphoblastic leukemia (ALL)

  * High-risk disease
* Participation in clinical trial COG-P9906 required (pilot project)

  * In complete remission
  * Consented to future studies using banked tissue specimens
* Participation in clinical trial and COG-AALL03B1 and linked therapeutic studies COG-AALL0232 and COG- AALL0331(expansion project)

  * Experienced a bone marrow relapse within 36 months of initial diagnosis
  * Consented to future studies using banked tissue specimens
  * Have matched ALL blast and germline specimens
  * Demographic, clinical and pathologic data elements for these biospecimens available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Targets for High-Risk Pediatric Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of regions of copy number abnormalities (CNA) and uniparental disomy in leukemic lymphoblasts using Affymetrix GeneChip Mapping 500K array sets
Identification of regions of CNA and loss-of-heterozygosity using Affymetrix SNP 6.0 microarrays. (Expansion project)
Gene expression profiles for leukemic lymphoblasts using Affymetrix U133 Plus 2.0 arrays
Global expression of microRNAs in leukemic lymphoblasts using microRNA gene chips
Epigenomic profiles using the HpaII tiny fragment Enrichment by Ligation-mediated PCR (HELP) assay. (Expansion project)
Prioritization of candidate genes and genomic regions for resequencing using array-generated gene expression data and data for CNAs
Identification of genes that are consistently mutated in leukemic lymphoblasts using high-throughput focused gene resequencing

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Hunger, MD, Study Chair — Children's Hospital Colorado Center for Cancer and Blood Disorders
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States